CLINICAL TRIAL: NCT02095015
Title: Mucopolysaccharidosis (MPS) I, II, and VI Screening in a High Risk Population With Previous Surgical Repair or Presence of Inguinal and/or Umbilical Hernia in Combination With Pediatric Ear, Nose and Throat (ENT) Surgery (Adenoidectomy and/or Tonsillectomy and/or Tympanostomy) (The HATT Project)
Brief Title: Mucopolysaccharidosis (MPS) I, II, and VI Screening in a High-Risk Population With Previous Surgical Repair or Presence of Inguinal and/or Umbilical Hernia in Combination With Pediatric ENT Surgery (The HATT Project)
Status: Terminated | Type: Observational
Why Stopped: terminated for not meeting enrollment goals
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SHP-001-801
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Mucopolysaccharidosis (MPS)
Keywords: MPS II; iduronate-2-sulfatase; Mucopolysaccharidosis VI; MPS; MPS VI; ear, nose and throat; Mucopolysaccharidosis II; Hunter syndrome; ENT; Mucopolysaccharidosis I; Hurler, Hurler-Scheie, or Scheie syndrome; Mucopolysaccharidosis; MPS I; Maroteaux-Lamy syndrome
MeSH Terms: conditions — Mucopolysaccharidoses; Sudden Infant Death; Mucopolysaccharidosis VI; Mucopolysaccharidosis II; Mucopolysaccharidosis I

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Analysis population: All subjects enrolled in the study who meet the eligibility criteria

SUMMARY:
Mucopolysaccharidosis (MPS) type II (MPS II; Hunter syndrome) is a rare, X-linked disease caused by a deficiency of the lysosomal enzyme iduronate-2-sulfatase (I2S) and occurs almost exclusively in boys, with an incidence of approximately 1.3 per 100,000 live male births.1 Early identification of MPS II is challenging because some initial features, such as chronic runny nose, otitis media, and hernias, are commonly seen in the general population. As a result, even though the signs and symptoms of MPS II typically appear early in childhood, the diagnosis may lag behind by several years.

The primary objective of this international multi-center study is to evaluate the positive screening rate of MPS II subjects by screening a high-risk male pediatric population who have had or are scheduled for 1 or more specific ENT surgical procedures (adenoidectomy and/or tonsillectomy and/or tympanostomy) and who have a previously repaired or present evidence of an inguinal and/or umbilical hernia.

DETAILED DESCRIPTION:
With evidence-based information from MPS registries regarding the types of surgical interventions that are most prevalent in MPS, this screening study is expected to provide the understanding of the role pediatric ENT surgeons can play in identifying young children with MPS.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet the following criteria to be enrolled in this study:

1. The subject is male.
2. The subject is <7 years of age.
3. The subject has had or is scheduled for ENT surgery for any of the following, alone or in combination: adenoidectomy, tonsillectomy, and tympanostomy.
4. The subject has record of previous surgical repair or presence of inguinal and/or umbilical hernia.
5. The subject's parent(s) or the subject's legally authorized representative(s) has provided written informed consent that has been approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC).

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. The subject has a current confirmed diagnosis of any MPS disorder.
2. The subject was born prematurely (defined as born before 37 weeks gestation).
3. The subject has received a blood transfusion within the past 6 weeks.
4. The subject has received a bone marrow transplant.

Max Age: 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Males of any ethnic background or race, <7 years of age or under, who have had or are scheduled for adenoidectomy and/or tonsillectomy and/or tympanostomy (alone or in combination), will be enrolled. In addition, the subjects must have previous surgical repair or presence of inguinal and/or umbilical hernia.
Sampling Method: Non-Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2014-05-21 (Actual); Primary Completion 2015-08-14 (Actual); Study Completion 2015-08-14 (Actual)

PRIMARY OUTCOMES:
The status of diagnosis of MPS II (either positive or negative) of each subject | Screening visit
  To evaluate the positive screening rate of MPS II subjects by screening a high risk male pediatric population.

SECONDARY OUTCOMES:
The status of diagnosis of MPS I or VI (either positive or negative) of each subject | Screening visit

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (14):
- United States (7):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Nemours Children's Clinic, Jacksonville, Florida
  - Children's Hospital and Clinic, Minneapolis, Minnesota
  - Saint Louis Children's Hospital, St Louis, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Intermountain Ear Nose and Throat Center, Salt Lake City, Utah
- Montreal Children's Hospital, Montreal, Quebec, Canada
- Italy (2):
  - Ospedale San Gerardo, Monza
  - Ospedale Pediatrico Bambino Gesù, Passoscuro
- Christus Muguerza del Parque, S.A. de C.V., Chihuahua City, Mexico
- Hospital de Cruces, Barakaldo, Spain
- Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara, Turkey (Türkiye)
- Royal Manchester Children's Hospital, Manchester, United Kingdom

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fd24db2bf003ab46abe